CLINICAL TRIAL: NCT05572021
Title: A Comparison of the Outcomes in Fortiva and Strattice Mesh
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00088523
Record Dates: First submitted 2022-10-06; First posted 2022-10-07 (Actual); Results first posted 2025-10-28 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2024-09

CONDITIONS: Ventral Hernia
Keywords: ventral hernia; surgical biologic mesh; hernia complications
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Intervention Model Description: Comparison of prospective group to retrospective group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Prospective (Experimental): Participants enrolled to ventral hernia repair with Fortiva mesh
  Interventions: Device: Prospective Ventral Hernia Repair with Fortiva
- Retrospective (Active Comparator): Retrospective participants with ventral hernia repair using Strattice mesh
  Interventions: Device: RetroSpective Ventral Hernia Repair with Strattice

INTERVENTIONS:
Device: Prospective Ventral Hernia Repair with Fortiva — Ventral hernia repair using Fortiva biologic mesh
  Arms: Prospective
Device: RetroSpective Ventral Hernia Repair with Strattice — Retrospective cohort of ventral hernia repair patients using Strattice mesh
  Arms: Retrospective

SUMMARY:
A comparison of ventral hernia repair with Strattice and Fortiva mesh.Primary The study team aims to determine the hernia recurrence rates for RTI Surgical biologic mesh (Fortiva) compared to Strattice. Also the study team aims to determine the mesh related complications for RTI Surgical biologic mesh (Fortiva) compared to Strattice

DETAILED DESCRIPTION:
This study will be a prospective, matched study of patients using Fortiva biologic mesh to determine the rates of hernia recurrence and mesh related complication compared to Strattice mesh. Patients who meet the inclusion and exclusion criteria will be prospectively enrolled to receive a Ventral Hernia Repair (VHR) using Fortiva biologic mesh and will be compared to a retrospective cohort of patients with a VHR that utilized Strattice mesh. Patients will be propensity matched in a 1:3 (Fortiva : Strattice) fashion based on age, sex, and hernia defect size.

ELIGIBILITY:
Inclusion Criteria:

* Ventral Hernia requiring surgical repair

Exclusion Criteria:

* Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-03-21 (Actual); Study Completion 2025-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Heniford, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Carolinas Medical Center, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study planned to use matched analysis matching the prospective and retrospective arms. For studies of this fashion all prospective participants are enrolled first to sample size and then matching retrospective patients are enrolled. It is not a standard practice to match patients as they enroll. This study was terminated before prospective arm enrollment was completed. Therefore, no participants were enrolled in the retrospective arm.
Period: Overall Study
Arm/Group | Prospective | Retrospective
Started | 6 | 0
Completed | 1 | 0
Not Completed | 5 | 0
Not completed — Study terminated - PI left the institution and no other surgeons were interested in continuing study | 5 | 0

BASELINE CHARACTERISTICS:
Population: This study planned to use matched analysis matching the prospective and retrospective arms. For studies of this fashion all prospective participants are enrolled first to sample size and then matching retrospective patients are enrolled. It is not a standard practice to match patients as they enroll. This study was terminated before prospective arm enrollment was completed. Therefore, no participants were enrolled in the retrospective arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prospective | Retrospective | Total
Number analyzed (Participants) | 6 | 0 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.0 (6.8) |  | 66.0 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 4
  Male | 2 |  | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 6 |  | 6
  Unknown or Not Reported | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 6 |  | 6
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Participants With a Hernia Recurrence
Description: Frequency of participants with a hernia recurrence
Time Frame: 1 year follow up post surgical repair
Population: as for baseline characteristics
Measure: Number; unit: occurrence
Arm/Group | Prospective | Retrospective
Number analyzed (Participants) | 1 | 0
occurrence | 0 |

2. Primary Outcome: Percentage of Participants With a Hernia Recurrence
Description: Percentage of participants with a hernia recurrence
Time Frame: 1 year follow up post surgical repair
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Prospective | Retrospective
Number analyzed (Participants) | 1 | 0
percentage of participants | 0 |

3. Secondary Outcome: Number of Participants With a Mesh Related Complication
Description: Number of participants with a mesh related complication
Time Frame: 1 year follow up post surgical repair
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Prospective | Retrospective
Number analyzed (Participants) | 1 | 0
Participants | 0 |

4. Secondary Outcome: Percent of Participants With a Mesh Related Complication
Description: Percent of participants with a mesh related complication
Time Frame: 1 year follow up post surgical repair
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | Prospective | Retrospective
Number analyzed (Participants) | 1 | 0
percentage of participants | 0 |

ADVERSE EVENTS:
Time Frame: Baseline through 6 months. After 6-months events were not attributed to surgical procedure.
Description: This study planned to use matched analysis matching the prospective and retrospective arms. For studies of this fashion all prospective participants are enrolled first to sample size and then matching retrospective patients are enrolled. It is not a standard practice to match patients as they enroll. This study was terminated before prospective arm enrollment was completed. Therefore, no participants were enrolled in the retrospective arm.
Arm/Group | Prospective | Retrospective
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/0
Other Adverse Events (participants affected / at risk) | 0/6 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-28): https://cdn.clinicaltrials.gov/large-docs/21/NCT05572021/Prot_SAP_001.pdf
  • Informed Consent Form (2025-05-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT05572021/ICF_000.pdf